CLINICAL TRIAL: NCT07358429
Title: Effects of CPAP Therapy on Atrial Fibrillation Recurrence in Patients With Obstructive Sleep Apnea: A Prospective Cohort Study
Brief Title: CPAP Therapy and Atrial Fibrillation Recurrence in OSA
Acronym: CPAP-AF
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Sofia (Other)
Responsible Party: Principal Investigator, Petar Rosenov Kalaydzhiev, Assistant Professor, Medical University of Sofia
Other Study IDs: MP18/09.08.2024
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea (OSA); Atrial Fibrillation (Paroxysmal)
Keywords: sleep apnea; atrial fibrillation; CPAP therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Atrial Fibrillation; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High CPAP adherence (≥ 4 h/night): Participants with mean nightly CPAP use ≥ 4 hours.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- Low CPAP adherence (< 4 h/night): Participants with mean nightly CPAP use < 4 hours.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — CPAP therapy is initiated according to standard clinical practice. Objective adherence data (mean nightly usage, percentage of nights ≥ 4 hours) are collected via telemonitoring systems.

SUMMARY:
Obstructive sleep apnea (OSA) is a major modifiable risk factor for atrial fibrillation (AF). Continuous positive airway pressure (CPAP) therapy has been shown to improve cardiovascular outcomes; however, real-world data on its effect on AF recurrence remain limited.

This prospective cohort study aims to evaluate the association between objective CPAP adherence and the risk of AF recurrence in patients with moderate-to-severe OSA and a history of paroxysmal AF.

Patients will be followed for 12 months, with AF recurrence assessed using electrocardiography and Holter monitoring.

DETAILED DESCRIPTION:
This is a prospective, real-world cohort study enrolling adult patients with moderate-to-severe obstructive sleep apnea (AHI ≥ 15 events/hour) and documented paroxysmal atrial fibrillation. OSA is diagnosed using home sleep apnea testing.

All participants initiate CPAP therapy, with objective adherence data collected via telemonitoring. Patients are followed for 12 months to assess AF recurrence, progression to permanent AF, and associations with CPAP usage metrics.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosed moderate-to-severe OSA
3. History of paroxysmal atrial fibrillation
4. Ability to initiate CPAP therapy
5. Written informed consent -

Exclusion Criteria:

1. Left ventricular ejection fraction < 50%
2. Permanent atrial fibrillation
3. Central sleep apnea
4. End-stage chronic kidney disease
5. Inability to obtain or tolerate CPAP therapy -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with moderate-to-severe obstructive sleep apnea and a history of paroxysmal atrial fibrillation, managed in outpatient and hospital settings, and treated with continuous positive airway pressure therapy as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to First Recurrence of Paroxysmal Atrial Fibrillation | 12 months
  First documented recurrence of paroxysmal AF confirmed by 12-lead ECG or 24-hour Holter monitoring.

SECONDARY OUTCOMES:
Progression to Permanent Atrial Fibrillation | 12 months
  Progression to Permanent Atrial Fibrillation for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Petar R Kalaydzhiev, PhD, Principal Investigator — Medical University - Sofia
Locations (1):
- UMHAT "Tcaritca Joanna - ISUL", Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to data protection regulations and the absence of explicit participant consent for data sharing beyond the scope of the current study.